CLINICAL TRIAL: NCT06291870
Title: Predictors of Post-COVID Clinical and Cognitive Consequences
Brief Title: Predictors of Post-COVID-19 Clinical and Cognitive Consequences
Acronym: SCLC
Status: Recruiting | Type: Observational
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: John D. Dingell VA Medical Center (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: F4396-P; IRB-22-01-4294 (Other: John D. Dingell VA Medical Center)
Record Dates: First submitted 2024-03-01; First posted 2024-03-04 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Post Acute Sequelae of SARS CoV 2 Infection; Obstructive Sleep Apnea
Keywords: COVID-19; Quality of Life; Neurocognitive Function; Sleepiness; Sleep Quality; Six minute walk; Fatigue
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome; Sleep Apnea, Obstructive; COVID-19; Sleepiness; Sleep Initiation and Maintenance Disorders; Fatigue

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Biospecimen Retention: Samples With DNA — blood ApoE
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- COVID+: Patients with post-acute sequelae of SARS-COV-2 infection (PSAC) and obstructive sleep apnea (OSA)
- Control: Patients with obstructive sleep apnea and no history of COVID-19

SUMMARY:
The CDC describes Post-acute sequelae of SARS-COV-2 infection (PASC) for the wide range of physical and mental health consequences experienced by some patients. These sequelae may be present four or more weeks after SARS-COV-2 infection, including patients who had initial mild or asymptomatic acute infection. However, there is complete absence of data whether chronic sleep changes due to COVID-19 infection may influence these physical and mental health consequences. While fatigue is one of the common post-COVID conditions, there are no systematic examinations of sleep disturbances in COVID-19 survivors. This will be a pilot observational retrospective and prospective cohort study, to systematically assess if sleep disturbances and severity of sleep apnea comprise a modifiable facet of PASC as well as the short-term and longer-term effects of COVID-19 infection itself on sleep, cognitive function, exercise capacity and lung function.

DETAILED DESCRIPTION:
This pilot study will systematically collect data to assess if sleep disturbances and severity of sleep apnea comprises a modifiable facet of PASC. This study will be the first step towards collecting preliminary data for a larger, longer-duration and more comprehensive study regarding the relationships between long-COVID and sleep disturbances which can inform future healthcare strategies and clinical decision-making. The study will also explore whether inflammatory biomarkers levels during acute COVID infection predict severity and duration of long-COVID or PASC and sleep fragmentation post-COVID.

Objectives: The overall goal of this project is to determine the associations between chronic post-COVID fatigue and sleep duration and sleep quality in patients after recovery from SARS-CoV-2 infection. The investigators have adopted the CDC definition for Post-COVID Conditions which persist for four or more weeks after SARS-CoV-2 infection and also is known as Post-Acute Sequelae of SARS-COV-2 infection (PASC).

Specific Aim 1: Determine associations between sleep duration and sleep quality on PASC-related fatigue symptoms, cognitive function, biomarker levels and vigilance.

Specific Aim 2. Determine if presence of obstructive sleep apnea (OSA) and level of PAP adherence during and prior to COVID-9 infection in patients with OSA predicts PASC- related fatigue, cognitive function and quality of life (QoL).

Exploratory Aim: Determine whether partial or full/booster vaccinations with COVID-19 mRNA vaccine vs. no vaccination has an impact on chronic post-COVID fatigue and sleep disturbances.

ELIGIBILITY:
Inclusion Criteria:

* All individuals 18 years or older, with prior history of COVID-19 infection diagnosis
* Both genders including all racial and ethnic groups
* Patients with OSA (apnea hypopnea index of 5/hour on polysomnography) with history of COVID-19 infection will be eligible with prior history of COVID-19 infection and without COVID-19 for Aim 2

Exclusion Criteria:

* Inability to give consent
* Active suicidal symptoms
* Children of all ages
* Pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The investigators will include all individuals 18 years or older, both genders, all racial and ethnic groups, with diagnosis of COVID-19 infection, diagnosed using any validated antigen detection test and/or polymerase chain reaction (PCR) test and of any severity level of COVID. Eligible patients with COVID-19 history of infection should be at least 1 month after the diagnosis of COVID-19 and should have been discharged to home if admitted to an acute care facility. COVID-19 antigen test positive patients who were completely asymptomatic at the time of COVID positive testing will be excluded. Controls will be patients without history of COVID-19 infection and age 18 years or older. In addition, patients with OSA (apnea hypopnea index = of 5/hour on polysomnography) with history of COVID-19 infection will be eligible for Aim 2.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-01-19 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Neurocognitive function Trails A and Trails B | Change from baseline at 3 months
  Trails A and Trails B test will be administered to evaluate attention and psychomotor function. This score is adjusted for age, race, gender, and years of education. Scored on a Standard scale of 100 +/- 15 for normal ranges, above 115 is above average, below 85 is considered below average.
Neurocognitive function PASAT | Change from baseline at 3 months
  PASAT (Paced Auditory Serial Addition Test) will be administered to evaluate vigilance and executive function. The PASAT is recorded as the total number of correct responses (from 0-60), or the percent of correct responses out of 60 (from 0-100), where a higher value is a better outcome.
Neurocognitive function Stroop color-word interference | Change from baseline at 3 months
  Stroop color-word interference test will be administered to evaluate executive function. This score is adjusted for age, and years of education. Scored on a Standard scale of 100 +/- 15 for normal ranges, above 115 is above average, below 85 is considered below average.
Neurocognitive function DIGIT | Change from baseline at 3 months
  DIGIT test will be administered to evaluate short-term and working memory. This score is adjusted for age. Scored on a Standard scale of 100 +/- 15 for normal ranges, above 115 is above average, below 85 is considered below average.
Neurocognitive function WASI | Change from baseline at 3 months
  Abbreviated Wechsler Abbreviated Scale of Intelligence (WASI) will be administered to evaluate verbal comprehension and working memory. This score is adjusted for age. Scored on a Standard scale of 100 +/- 15 for normal ranges, above 115 is above average, below 85 is considered below average.
Neurocognitive function WMS | Change from baseline at 3 months
  Wechsler Memory test (WMS) will be administered to measure Verbal comprehension, and working and visual memory. Scored on a Standard scale of 100 +/- 15, where a higher score is a better outcome.
Neurocognitive function PVT | Change from baseline at 3 months
  Psychomotor Vigilance Test (PVT) will be administered to measure Alertness and vigilance, in terms of number of lapses and reaction time. The performance score ranges from 0-100, where a higher value is a better outcome.
Neurocognitive function HVLT-R | Change from baseline at 3 months
  Hopkins Verbal Learning Test - Revised (HVLT-R) will be administered to evaluate Verbal learning and memory. Scored on a Standard scale of 100 +/- 15, where a higher score is a better outcome.
Sleepiness ESS | Change from baseline at 3 months
  Epworth sleepiness scale (ESS) score will be measured. This score is on a scale of 0-24, where a higher value indicates greater degree of sleepiness.
Sleep quality PSQI | Change from baseline at 3 months
  Pittsburgh Sleep Quality Index (PSQI) is a detailed assessment of subject sleep quality over the most recent month by considering seven "component" scores: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleeping medication, and daytime dysfunction. The sum of scores for these seven components yields one global score to assess sleep quality on a scale of "poor" to "good".
Quality of life SF-36v2 | Change from baseline at 3 months
  QoL will be assessed using the survey SF-36v2 Health survey. Thirty-five of the SF-36v2 items are used to measure eight domains of health-related quality of life. These are on a scale of 0-100, where higher values indicate a better outcome.
Quality of life FOSQ | Change from baseline at 3 months
  Disease specific QoL will be assessed using the Functional Outcomes of Sleep Questionnaire FOSQ/(FOSQ). There are 5 subscale domains of the FOSQ (General Productivity, Social Outcome, Activity Level, Vigilance, and Intimate Relationships and Sexual Activity). There all range from 0-20, where a higher value is a better outcome. The total FOSQ is the sum of these subscale domains and ranges from 0-100, where a higher value is a better outcome.
Quality of life SGRQ | Change from baseline at 3 months
  Disease specific QoL will be assessed using the St. George's Respiratory Questionnaire (SGRQ). The SGRQ has three subscale domains (Symptoms, Activity, and Impacts), which range from 0-100, where a higher value indicates a worse outcome. The total SGRQ is the average of these subscale domains and is on a scale of 0-100, where a higher value is a worse outcome.
Fatigue Severity | Change from baseline at 3 months
  Fatigue Severity Scale (FSS): FSS measures how fatigue affects motivation, exercise, physical functioning, carrying out duties, interfering with work, family, or social life. Where a higher value is a worse outcome.
PROMISE Sleep Disturbance | Change from baseline at 3 months
  Sleep disturbance short form assesses sleep disturbance over the past seven days.
Horne and Osteberg Morningness/Eveningness Questionnaire | Change from baseline at 3 months
  Morningness/Eveningness Questionnaire measures the degree of which respondents are active and alert at certain times of the day. Scale is 1 to 5.
Mini Mental State Examination (MMSE) | Change from baseline at 3 months
  Mini Mental State Examination (MMSE) is a simple way to quantify cognitive function and screen for cognitive loss. This score is on a scale of 0-30, a larger value is a better outcome.
Borg Scale | Change from baseline at 3 months
  This measures the level of dyspnea during the 6 minute walk test. It is on a scale of 0-10, where a larger value is a worse outcome.
Dyspnea: Six-minute walk test (6MWT) distance | Change from baseline at 3 months
  Participants are instructed to achieve maximal distance. There is no scale, but a larger value is a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Susmita Chowdhuri, MD MS, Principal Investigator — John D. Dingell VA Medical Center, Detroit, MI
Locations (1):
- John D. Dingell VA Medical Center, Detroit, MI, Detroit, Michigan, United States

IPD SHARING:
Plan to Share IPD: No